CLINICAL TRIAL: NCT06641154
Title: A Phase I/II, Open Label, Study to Evaluate Safety and Efficacy of an Intravenous Injection of GT-UGT1A1-AAV8-02 (AAV Vector Expressing the UGT1A1 Transgene) in Patients with Crigler-Najjar Syndrome Type I Requiring Phototherapy
Brief Title: Gene Therapy for Crigler Najjar Syndrome Type I (AlphaCN)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Federal State Budget Institution Research Center for Obstetrics, Gynecology and Perinatology Ministry of Healthcare (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GT-UGT1A1-AAV8-02
Record Dates: First submitted 2024-10-11; First posted 2024-10-15 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2024-11

CONDITIONS: Crigler-Najjar Syndrome Type I
Keywords: Crigler-Najjar syndrome type I; gene therapy; GT-UGT1A1-AAV8-02; Adeno Associated Virus; Crigler-Najjar
MeSH Terms: conditions — Crigler-Najjar Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- GT-UGT1A1-AAV8-02 (Experimental): 2 doses of the IMP assessed in the dose escalation, open-label, phase 1/2 study
  Interventions: Drug: GT-UGT1A1-AAV8-02

INTERVENTIONS:
Drug: GT-UGT1A1-AAV8-02 — Intravenous infusion, single dose
  Other Names: alphaglucuronosyltransferasegene unoparvovec; alphacrigen; OGP-001; AAV-TBG1A1

SUMMARY:
This is a Phase 1/2, multinational, open-label, study to evaluate the safety and efficacy of an intravenous infusion of GT-UGT1A1-AAV8-02 in patients with Crigler-Najjar type 1 aged ≤10 years and requiring phototherapy. Patients will received a single administration of GT-UGT1A1-AAV8-02 and will be followed for safety and efficacy of approximately 60 months (5 years):

* a follow-up of approximately 12 months (48 weeks)
* a long term follow-up of approximately 48 months (4 years), in order to be in line with the latest EMEA Guideline on follow-up of patients administered with gene therapy medicinal products, released on 22 Oct.2009 by the Committee for medicinal products for human use.

DETAILED DESCRIPTION:
Inherited enzymopathy of uridine diphosphate glucuronosyltransferase 1A1 (Crigler-Najjar syndrome type I) is an orphan disease, that arises from loss of function UGT1A1 genetic variants. Mutations lead to the enzyme's inability in neutralization of bilirubin conjugates. Clinically this condition is represented by jaundice and severe neurologic disorders, which can lead to death in infancy. Diagnosis of Crigler-Najjar syndrome type I is made through biochemical tests and determination the level of unconjugated bilirubin in blood serum, as well as by molecular genetic methods. There is no specific treatment for the disease, except liver transplantation. In common clinical practice phototherapy and plasmapheresis are applied in order to reduce serum concentration of unconjugated bilirubin and destroy or eliminate it from the body. From the very newborn and further, the lifestyle of young patients is dramatically restricted by the long-lasting exposure to phototherapy.

In Russian Federation there are just a few children annually with such disorder. Under our vision is a girl diagnosed Crigler-Najjar type I, who had either opportunity of liver transplantation and long term immunosuppression or receive a gene therapy within previously promising reports in clinics.

The Crigler-Najar syndrome is a convenient subject of choice for a gene therapy application, because the product of the damaged gene is directly related to a well-studied metabolite in the human body. The norms of bilirubin are known to biochemists, and it is clear how to study it's concentration in plasma. In addition, the level of bilirubin usually correlates well with the levels of liver enzymes, which reflect the condition of the liver and the possible viral load of gene constructs that have liver tropism.

Previously successful applications of gene therapy for this syndrome encouraged us to implement this treatment for the first time on children.

GT-UGT1A1-AAV8-02 (alphaglucuronosyltransferasegene unoparvovec, alphacrigen, OGP-001, AAV-TBG1A1) is comprised of a recombinant adeno-associated virus type 2/8 (rAAV2/8), carrying the normal human UGT1A1 gene. rAAV2/8 does not contain viral genes, but only viral inverted terminal repeats (ITRs), that are essential for genome rescue, replication, packaging, and vector persistence. Instead of viral genes, the vector carries a genetic engineering construct that ensures expression of the human UGT1A1 gene under the control of liver specific promoter of the human thyroxine-binding globulin (TBG) gene.

ELIGIBILITY:
Inclusion Criteria:

Patients with severe Crigler-Najjar syndrome resulting from a molecular confirmation of mutations in the UGT1A1 gene and requiring phototherapy male or female at least 3 months (no more 10 years) at the date of signature of informed consent Patient able to give informed assent and/or consent in writing

Exclusion Criteria:

Patients who underwent liver transplantation Patients with chronic hepatitis B or C Patients infected with Human immunodeficiency virus (HIV) Patients with significant underlying liver disease Patients with significant encephalopathy Participation in any other investigational trial during this trial Patients unable or unwilling to comply with the protocol requirements

Ages: 3 Months to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 5 (Estimated)
Dates: Start 2024-11-06 (Actual); Primary Completion 2027-11-01 (Estimated); Study Completion 2029-11-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients having received the selected dose of GT-UGT1A1-AAV8-02 with serum bilirubin ≤ 300µmol/L within 48 meeks after GT-UGT1A1-AAV8-02 administration and without phototherapy from week 16 | 48 weeks
  Decrease of total Serum bilirubin level after interruption of daily phototherapy (Efficacy); change in serum total biliirubin from baseline to week 48
Incidence of Treatment Emergent Adverse Events or Treatement Serious Adverse Events | 48 weeks
  Incidence of AE/SAE evaluated by changes in laboratory parameters, vital signs, physical examination, reported from baseline to each visit study. Clinically relevant abnormal findings on Laboratory values, Vital Signs, Physical findings will be reported as Adverse Events.
  Incidence and Severity of Adverse Events for each body system will be presented for each dose level and summarized overall.

SECONDARY OUTCOMES:
Change in Health-related quality of Life for Children from Baseline to Week 48 after GT-UGT1A1-AAV8-02 administration | 48 weeks
  Quality of Life outcome measure: change of quality of life from Baseline to Week 48 after GT-UGT1A1-AAV8-02 administration.
  PedsQL 4.0 Generic Core Scale for pediatrics: 0-100 scale where higher scores indicate better health-related quality of life

CONTACTS AND LOCATIONS:
Locations (2):
- Russia (2):
  - Alphaviva LLC, Moscow
  - Federal State Budget Institution Research Center for Obstetrics, Gynecology and Perinatology Ministry of Healthcare, Moscow

IPD SHARING:
Plan to Share IPD: Undecided